CLINICAL TRIAL: NCT03422614
Title: Pathophysiologie Angeborener Immundefekte
Brief Title: Pathophysiology of Inborn Immunodeficiencies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Janine Reichenbach, Co-Head Division Immunology, University of Zurich
Other Study IDs: Patho_PID
Record Dates: First submitted 2018-01-10; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients with Primary Immunodeficiency
  Interventions: Diagnostic Test: Diagnostic Test
- Control: Healthy Controls
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Characterisation of cellular and functional phenotype in different PIDs

SUMMARY:
The pathophysiology of primary immunodeficiencies (PID), which encompass a broad range of different diseases with susceptibility to infection and/or a deregulated inflammatory response, is poorly understood. Available treatments are often not specific for a distinct target and might be associated with side effects. To elucidate pathophysiology of different PIDs, stool, urine, blood, tissue biopsies and/or bone marrow will be collected and analysed for anti-microbial activity and inflammatory response. In a second step, targeted treatment for different PIDs might be developed preclinically and ex vivo according to underlying pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an inborn error of immunity (primary immunodeficiency, PID)
* Clinically healthy (non-age matched) volunteer

Exclusion Criteria:

* exclusion of an inborn error of immunity
* secondary immunodeficiency
* refusal to enter the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PID and healthy controls of all ages might be tested, recruitment is in a tertiary care hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterisation of cellular phenotype in different PIDs | immediately after sampling of biological specimen or up to 10 years later from frozen samples
  Immune cell subsets will be analysed for Surface marker Expression or cell activation pathways
Characterisation of functional phenotype in different PIDs | immediately after sampling of biological specimen or up to 10 years later from frozen samples
  Immune cell subsets will be analysed for cytokine production or cell activation pathways

SECONDARY OUTCOMES:
Identification of potential targets for pathophysiology-specific treatment, or for curative treatment such as gene therapy for different PIDs ex vivo | immediately after sampling of biological specimen or up to 10 years later from frozen samples
  Targets for development of new Treatment for PID identfied by Primary outcome analyses (see above) can be pathways, Surface marker Expression or cytokine production. Therefore new Treatment developed might consist of medication interfering with cell activation pathways, cytokine production (e.g. inhibitory antibodies against specific cytokines) or Surface marker Expression (e.g. inhibitory or stimulatory ligands for certain cell Surface receptors)

CONTACTS AND LOCATIONS:
Overall Officials: Janine Reichenbach, Prof. Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share IPD in the form of Scientific publications in peer-reveiwed journals and communications at Scientific meetings